CLINICAL TRIAL: NCT04537585
Title: A Multi-center, Investigator-blinded, Randomized Clinical Trial, 18-months, Parallel-group to Compare the Efficacy of Tomeka® Foods Versus Vernonia Amygdalina in the Prevention and Maintenance of Remission of COVID-19 in DRC
Brief Title: COVID-19: Collecting Measurements of Renin-angiotensin-system Markers, Such as Angiotensin-2 and Angiotensin 1-7
Acronym: Tomeka
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guyguy K Tshima, MD (Other)
Collaborators: Centre Médical de Kinshasa (CMK) (Unknown)
Responsible Party: Sponsor-Investigator, Guyguy K Tshima, MD, Coordinator, University of Kinshasa
Organization: University of Kinshasa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TOMEKA
Record Dates: First submitted 2020-08-29; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: Covid 19; Tomeka®; Vernonia amygdalina; Selenium; DRC
MeSH Terms: conditions — COVID-19 | interventions — MAZE protocol; Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Investigators couldn't agree more to wait without to know how to treat their patients better and want to learn about therapeutic nutrition approach called TOMEKA versus prophylaxis dosing of antioxidant as Vernonia amygdalina as a study. Investigators are learning about that here in September, why wasn't that done in April? Investigators would submit to follow a parallel group, just speaking as researchers about randomisation, one of the reasons difficult to reach that elaborate study design is sometimes bureaucracy is just daunting.
Masking Description: The fact that you can't really study anything unless there's funding for it because the insurance companies and the hospitals are not going to pay for things on a trial unless there is funding. Then you add to that there is no funding for food as medicine, and things as herbs like Vernonia amygdalina that improve the quality of life in COVID-19 patients and they are not pharmaceutical. Those are sort of the real-world complaints, investigators would say, on the front lines to follow participants in parallel group i.e. compare the ones who take herbs as medicine for their survival and other who use others means to fight COVID-19 symptoms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tomeka (Experimental): Number of participants with treatment-TOMEKA® usage as assessed by Education [ Time Frame: 18 months ] Change people's behaviour
  Interventions: Combination Product: Tomeka®; Drug: "Vernonia amygdalina"
- "Vernonia amygdalina" (Experimental): Number of participants with "Vernonia amygdalina" herbs usage as assessed by Education [ Time Frame: 18 months ] Change people's behaviour
  Interventions: Combination Product: Tomeka®; Drug: "Vernonia amygdalina"

INTERVENTIONS:
Combination Product: Tomeka® — Tomeka® is a farine mixte made by soy, sorghum, maze and mushrooms
  Other Names: Maze; Soy; Sorghum; Mushrooms
Drug: "Vernonia amygdalina" — "Vernonia amygdalina" is the Intervention that was pre-specified to be administered as part of the protocol as a particular intervention of not "of interest" because the World Health Organization doesn't support its use due to two reports case of toxicity in Kinshasa in a child and Mbandaka in an adult in the Democratic Republic of the Congo that why investigators would like review its usage in a large community and update that intervention of not "of interest" as appropriate (using randomisation on the follow up of participants who will take by themselves those herbs called Congo Bololo to compare, as necessary, to the ones who are afraid to take them because of reported cases of toxicity).
  Other Names: Congo Bololo (D. R. Congo); grawa (Amharic); ewuro (Yoruba); etidot (Efik); onugbu (Igbo); ityuna (Tiv),; oriwo (Edo); Awɔnwono (Akan); chusar-doki (Hausa),

SUMMARY:
Investigators study meet the World Health Organization definition of a clinical trial because it is a prospective study in which participants will be assigned to intervention groups to investigate the effects on health outcomes. Investigators highlighted clearly the real problem that indigeneous patients are facing now in the Democratic Republic of the Congo: Poverty meaning the lack of money to buy goods and drugs. From the news report, investigators learned that "In the Democratic Republic of the Congo, indigenous communities in Kananga, Tshikapa and in the Kasai region are increasing their consumption of "Vernonia amygdalina," a traditional plant believed to cure several diseases, including alleviating COVID-19." Based on an unpublished work, quite a few extract molecules of Vernonia amygdalina are excellent antiviral candidates which are the family members of Remdesivir in terms of their antiviral mechanisms. Furthermore, the antiviral capabilities of these molecules are significantly stronger than or at least equivalent to Remdesivir. The target zones of these molecules in the human body cover a set of important organs and tissues. For example, Vernolide (C19H22O7) is able to reside firmly at bronchi, the upper respiratory tract, and blood vessels.

From the news report, investigators learned also that Herbs used in Tanzania include lemon, ginger, neem tree leaves, mango tree leaves, orange tree leaves. These traditional medicines contain, more or less, antiviral molecules whose capacities range from good to outstanding levels. Those herbs have been used worldwide to fight COVID-19.

In conclusion traditional medicines have been playing important roles not only in Africa but also in Asia, in South America, etc. Herbs prove themselves with effective efficacies in many therapeutic practices.

So maybe after careful considerations, the World Health Organization may support the use of herbs for poor patients who cannot afford modern drugs and used traditional medicines after a positive COVID-19 test in the Democratic Republic of the Congo. Investigators are talking about a randomisation's nuance process to follow participants who decide by themselves if diagnosed positive to COVID-19 to begin to take herbs not waiting for a physician prescription.

DETAILED DESCRIPTION:
Background Selenium supplementation is suggested for an intervention better in food intake. The Tomeka Prevention Trial (TPT) is a randomized double blind nutri prevention trial. Initial blood collection will be specifically for the analysis of Selenium [antioxidant] and storage of serum. An additional blood collection will be carried out using anticoagulants so that plasma and white blood cells can be isolated. Plasma will allow the analysis of additional biomarkers collecting measurements of renin-angiotensin-system markers such as Angiotensin-2 and Angiotensin 1-7. This serum will be used (among other possible uses) for studies to investigate the antioxidant effect of Vernonia amygdalina in organs which may influence COVID-19 risk in emergency situations.

The TOMEKA WBC [white blood cell] sample will be available to TOMEKA investigators as well as outside researchers who have important, timely hypotheses to test. Because the sample bank is a limited resource, proposals to use it will be evaluated in terms of scientific relevance, significance, and validity as well as the potential impact of the proposed study. The amount and type of material needed will also be considered and the efficient use of material will be required. Strict confidentiality will be exercised and the information provided to investigators will not contain personal identifiers.

When specific uses of the TOMEKA WBC samples will be approved, the protocol will be amended.

Objectives To provide a resource for studies of early markers, etiology, and genetic risk factors for COVID-19. To collect measurements of renin-angiotensin-system markers, such as angiotensin-2 and angiotensin 1-7.

Methods Because the original model consent form did not specifically address herbal studies, participants will be asked to sign an additional consent form to document their consent to the collection and submission of additional blood samples for storage and future testing (including laboratory analysis). WHO? Everyone aged 15 and up experiencing symptoms of fever, cough, or shortness of breath with confirmed active COVID-19. WHY? To see if the investigational use of Tomeka® will prevent hospitalization and death, in COVID-19 patients. WHAT? The study type is observational after using patient individual data and investigators are assigned prospectively to monitor symptoms of the COVID-19 with a questionnaire. At the slightest symptom associated with the COVID-19 virus present in the patient's individual data, namely: fever (38 degrees c or 100, 4 degrees F), new or exacerbated cough, shortness of breath, sore throat, loss of smell, sudden onset without nasal congestion or loss of taste, digestive symptoms (nausea, vomiting / diarrhea), general weakness, headache, myalgia. Participants from the patient individual database will be randomized (like flipping a coin) to one of two groups. The intervention is education that needs to be evaluated with the suggested Tomeka® foods (nutraceuticals).

Conclusion The protocol presents a treatment model developed in its early stages with individual medical files. The principal investigator had the idea to create a treatment build or based on the principle of antioxidant supplementation, proteins, lipids, energy intake. The protocol is leading to a serious need of nutraceuticals solution faced to the missing cheap COVID-19 vaccine problem when it will be available. The nutritional status of each COVID-19-infected patient should be assessed prior to undertaking treatments. The outcome objective is to teach. The total budget required for the project is from 250.000 US$ to 1.000.000 US$ for education based on individual patient data and implementation on a global scale. This theoretical study merits further investigation for possible inclusion of nutraceuticals as an alternative for fighting and eradicating COVID-19.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for the trial must comply with all of the following at randomization:

1. Age ≥15 years
2. Current admission under the care of the heart-failure service at the site
3. Fulfill Inclusion criteria and accept
4. COVID-19 patients confirmed
5. be regular on appointments
6. No voluntary patient (see: having signed the informed consent) The criteria for choosing subjects: subjects who are themselves exposed to the consumption of Vernonia amygdalina (Kananga, Tshikapa or in Kasaï region). This group can be part of the cohort. tare: to compare with a no exposure group which is external to the cohort.

Here is the follow-up procedure for the two groups throughout the study:

* follow-up modality: visits, letters, work-study
* frequency of contacts: monthly
* total duration of follow-up: 9 months Patients enrolled in the individual data investigational study are potential candidates for TOMEKA intervention. As the TOMEKA protocol does not involve any investigational agents or techniques, patients would be eligible for dual randomization if they are themselves on stable doses of Vernonia amygdalina (the investigational herbs drugs may equivalent to Remdesivir).

Exclusion Criteria:

1. COVID-19 suspected clinically
2. Children
3. Refuse to participate
4. Recover when possible the cause of a study exit:

   * refusal of follow-up
   * move
   * death If the patient is no longer followed in the study without any cause being identified, then he is lost to follow-up.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-TOMEKA® usage | 18 months
  process assessed by Education

SECONDARY OUTCOMES:
Change From Baseline in herbs Vernonia amygdalina usage | 18 months
  take care of the Covid-19

CONTACTS AND LOCATIONS:
Overall Officials: Guyguy K. Tshima, MD, Principal Investigator — University of Kinshasa
Locations (1):
- Cliniques Universitaires de Kinshasa, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
The main thing investigators touched upon was funding, and they guess they would say that other researchers will frankly admit that they think just in terms of Food and herbs there are no funds for clinical trials. It will be through free websites that investigators plan to share their research. Mainly investigators plan to use Researchgate to share their results, also through peer-review journals and books.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18 months
Access Criteria: For free
URL: https://covind.org/

REFERENCES:
- Available data/document: Clinical Study Report: guyguytshimakabundi@gmail.com — http://cancovid.slack.com — It is a case of a baby from a COVID-9 positive mother who had a urogenital infection in the last two weeks of pregnancy. After the usual inflammatory assessment, investigators concluded that he had NEONATAL INFECTION, and put him on a triple combination of antibiotics (cefotaxime-clamoxyl-Gentamicin). On Day 3, the evolution was marked by a slight abdominal bloating, with a suspicion of a BEGINNING ULCERONECROSAN ENTEROCOLITIS and motivate the addition of Flagyl. On Day 4, the mother's anti-COVID serology came back positive and the father was also positive that motivated testing baby. Maybe the Covid-19 test was positive, investigators continued the same therapeutic regimen until Day 10; without the gentamicin that investigators had given for 5 days. On Day 10, the baby was asymptomatic. The baby was born by cesarean section indicated for scarring uterus. Free access data on demand. Review Board approval was required by the investigators by the time patient recruitment begins.